CLINICAL TRIAL: NCT04736836
Title: Rifaximin and Its Microbial Resistance as a Secondary Prophylaxis of Hepatic Encephalopathy in Patients With HCV Related Cirrhosis
Brief Title: Microbial Resistance of Rifaximin in Hepatic Encephalopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, Doaa abdelaziz, Part-Time Lecturer of pharmacy practice & clinical Pharmacy at Future University in Egypt, National Hepatology & Tropical Medicine Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CL(1173)
Record Dates: First submitted 2021-01-21; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- interventional (Active Comparator): 50 patient take rifaximin plus lactulose for 6 months
  Interventions: Drug: Rifaximin
- control (Placebo Comparator): 50 patient take lactulose for 6 months
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — locally absorbed antibiotic

SUMMARY:
Aims and Objectives: To determine the safety and efficacy of rifaximin plus lactulose as secondary prophylaxis of HE compared to lactulose alone. To evaluate the effect of long-term administration of rifaximin on development of resistant mutants and investigating its correlation with its efficacy.

Methods: An open label parallel, prospective interventional study was conducted. One hundred patients experienced at least one attack of hepatic encephalopathy were included in the study. Patients were randomly allocated either to receive rifaximin plus lactulose or lactulose alone for 6 months. Conn score, Model of End stage Liver Disease (MELD) score, asterixis grade, complete blood count (CBC), liver function tests, kidney function tests, urine and stool analysis and abdominal ultrasonography were compared in both groups. The primary efficacy endpoint was the time to the first breakthrough. The secondary efficacy endpoint was the time to the first hospitalization involving HE. Safety assessment was done by reporting any adverse events, serious adverse events and by repeating biochemical evaluation every 2 weeks. Determination of the minimum inhibitory concentration (MIC) of rifaximin for lactose fermenter isolates was done for the entire patients before starting treatment and at the end of treatment.

DETAILED DESCRIPTION:
Methodology Inclusion and exclusion criteria Fully conscious patients were enrolled from the National Hepatology and Tropical Medicine Research Institute (NHTMRI), Cairo, Egypt between January 2015 and December 2018. The inclusion criteria were cirrhosis due to HCV infection, age 18 to 75 years, experiencing at least one episode of OHE, and a MELD score ≤ 25.13 Patients with neurological or communication problems, hepatocellular carcinoma, diabetes mellitus, active infection, serum creatinine > 2 mg/dl, Hg < 8 g/dL, serum Na < 125 mmol/L or serum K < 2.5 mmol/L were excluded. Patients with previous intake of rifaximin as prophylaxis or any antibiotic within the last month were also excluded.

Study Design The protocol of this open label, parallel, prospective interventional study was approved by the institutional review board (IRB) of NHTMRI and that of the Faculty of Pharmacy, Cairo University (CL(1173)). All patients and/or patients' caregivers for those with weak/impaired cognitive and/or thinking ability due to previous episode of HE were consulted and explained for provided written informed consent before study enrolment.

The patients were randomly assigned into either intervention group (rifaximin group) or control group (lactulose only group). Both groups received lactulose syrup 30-45 ml three times daily while rifaximin 400 mg three times daily was added to the intervention group for 6 months. Other conventional therapy including diuretics, proton pump inhibitors, ursodeoxycholic acid and silymarin were given to the patients in both groups according to the hospital protocol.

Study Follow-up All recruited patients were assessed clinically and biochemically at baseline and every 2 weeks for 6 months. Conn score, asterixis grade, complete blood picture with differential, serum bilirubin (total and direct), serum aspartate transaminase (AST) and alanine transaminase (ALT), alkaline phosphatase, gamma-glutamyltransferase (GGT), serum albumin, prothrombin time and concentration, urea and serum creatinine, serum sodium (Na) and potassium (K), urine and stool analysis were measured.

Efficacy outcomes The primary efficacy endpoint was the time to the first breakthrough episode of OHE (defined as the time from the first dose of the study drug to an increase from a baseline Conn score of 0 or 1 to a score of 2 or more or from a baseline Conn score of 0 to a Conn score of 1 plus a 1-unit increase in the asterixis grade.13 The secondary efficacy endpoint was the time to the first hospitalization involving HE (defined as hospitalization because of the disorder or hospitalization during which an episode of HE occurred).14 The percentage of patient's survival during the study was also considered a secondary outcome.

Safety Outcomes All recruited patients were requested to report any adverse event(s) experienced during the study period. Clinic visits occurred every 2 weeks till end of the treatment period. On weeks with no clinical visits, patients were followed-up by phone calls.

Rifaximin Microbial Resistance Isolation of Gram negative bacteria from clinical stool samples Stool samples were collected from all the participants before commencing treatment and at the end of the study. One gram of stool was suspended in 10 ml saline and vortexed vigorously. One ml aliquot of the stool suspension was streaked on the surface of MacConkey agar plates to isolate Gram-negative lactose-fermenters. The plates were then incubated at 37⁰C for 24 hours. Pink colonies were picked and re-streaked one more time then suspended in 30% glycerol (vol/vol) in Brain Heart Infusion broth (BHI) and stored at -80 ⁰C till further analyses.

Determination of the minimum inhibitory concentration (MIC) of rifaximin for lactose fermenter isolates A sequential two-fold serial dilution broth procedure was adopted according to the Clinical and Laboratory Standards Institute (CLSI) guidelines.15 Ten dilutions of rifaximin were prepared starting from 256 μg/ml in Muller Hinton broth (MHB) and aliquoted in 200 μl aliquots in the wells of a round bottom 96-well plate. A control well was included that was prepared using 200 μl MHB inoculated with 20 μl of the prepared bacterial inoculum.

The inoculum was prepared by adjusting cells from an overnight culture to match the McFarland standard 0.5 (OD600 = 0.125). The suspension was further diluted 1:20 in MHB and 20 μl of the adjusted inoculum were added to each well. The plates were then incubated at 37°C for 24 hours. The experiment was repeated twice and the lowest concentration of rifaximin that resulted in complete inhibition of visible growth represented the MIC value. The MIC values were considered different if they differed by more than a two-fold dilution.16

ELIGIBILITY:
Inclusion Criteria:

- The inclusion criteria

1. cirrhosis due to HCV infection
2. age 18 to 75 years,
3. experiencing at least one episode of OHE,
4. MELD score ≤ 25

Exclusion Criteria:

1. Patients with neurological or communication problems,
2. hepatocellular carcinoma
3. diabetes mellitus
4. active infection
5. serum creatinine > 2 mg/dl, Hg < 8 g/dL, serum Na < 125 mmol/L or serum K < 2.5 mmol/L .
6. Patients with previous intake of rifaximin as prophylaxis or any antibiotic within the last month

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
the time to the first breakthrough episode of OHE the time to the first breakthrough episode of OHE (overt hepatic encephalopathy) | 6 months
  (defined as the time from the first dose of the study drug to an increase from a baseline Conn score of 0 or 1 to a score of 2 or more or from a baseline Conn score of 0 to a Conn score of 1 plus a 1-unit increase in the asterixis grade.

REFERENCES:
- [Derived] Zacharias HD, Kamel F, Tan J, Kimer N, Gluud LL, Morgan MY. Rifaximin for prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD011585. doi: 10.1002/14651858.CD011585.pub2. PMID 37467180
- [Derived] Abdel Moneim M, Abdelaziz DH, Ibrahim Nagy Y, Abdel Baki A, Attia AS, Sabry N. Rifaximin microbial resistance and its efficacy and safety as a secondary prophylaxis of hepatic encephalopathy in patients with hepatitis C virus-related cirrhosis. Int J Clin Pract. 2021 Nov;75(11):e14807. doi: 10.1111/ijcp.14807. Epub 2021 Sep 17. PMID 34487412